CLINICAL TRIAL: NCT00876460
Title: A Phase I Study of Continuous, Concomitant Oral Treatment With BIBF 1120 and Docetaxel - a Phase I, Open-label, Dose-escalation Study in Japanese Patients With Stage IIIB/IV or Recurrent Non-small-cell Lung Cancer After Failure of Chemotherapy
Brief Title: BIBF 1120 + Docetaxel (Japan) in Patients With Advanced Non-small-cell Lung Cancer, Phase I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1199.29
Record Dates: First submitted 2009-03-03; First posted 2009-04-06 (Estimated); Results first posted 2014-12-04 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

ARMS (1):
- BIBF 1120 + docetaxel (Experimental): Low, medium and high dose of BIBF 1120 and 60 mg/m2, 75 mg/m2 docetaxel every 3 weeks
  Interventions: Drug: BIBF 1120 M + docetaxel M; Drug: BIBF 1120 M + docetaxel H; Drug: BIBF 1120 H + docetaxel H; Drug: BIBF 1120 L + docetaxel M; Drug: BIBF 1120 H + docetaxel M

INTERVENTIONS:
Drug: BIBF 1120 M + docetaxel M — BIBF 1120 Medium dose bid + docetaxel 60 mg/m2
Drug: BIBF 1120 M + docetaxel H — BIBF 1120 Medium dose bid + docetaxel 75mg/m2
Drug: BIBF 1120 H + docetaxel H — BIBF 1120 HIgh dose bid + docetaxel 75 mg/m2
Drug: BIBF 1120 L + docetaxel M — BIBF 1120 Low dose bid + docetaxel 60 mg/m2
Drug: BIBF 1120 H + docetaxel M — BIBF 1120 HIgh dose bid + docetaxel 60 mg/m2

SUMMARY:
To confirm the safety of BIBF 1120 at a dose level up to 200 mg x 2/day (i.e., overseas recommended Phase III dose for combination treatment) with standard therapy of docetaxel (60 mg/m2 and 75 mg/m2) in Japanese advanced non small cell lung cancer (NSCLC) patients with stage IIIB/IV or recurrent after failure of first line chemotherapy and to determine the recommended dose for the Phase II trial.

ELIGIBILITY:
Inclusion criteria:

1. Histologically/cytologically confirmed, locally advanced/metastatic NSCLC of stage IIIB/IV or recurrent NSCLC (all histologies. Existence or nonexistence of measurable lesion according to RECIST is no object.)
2. Patients with one prior chemotherapy regimen including platinum-containing drug.

   In case of recurrent disease, one additional prior regimen is allowed for adjuvant and/or neoadjuvant therapy. However monotherapy of EGFR-TKI (i.e. erlotinib/Tarceva® and gefitinib/Iressa®) is not counted as 'one regimen'.
3. Male or female patients age >=20 years and =<74 years at the enrolment.
4. Life expectancy of at least three (3) months after the start of administration of the investigational drug.
5. Eastern Cooperative Oncology Group (ECOG) [R01-0787] performance Score 0 or 1.
6. Patients retaining a significant physiological compensatory function and patients with sufficient baseline organ function as follows:

   * Haemoglobin count more than 9.0g/dL
   * Absolute neutrophil count more than 1500/mm3
   * Platelet count more than 100 000/mm3
   * Serum creatinine less than or equal to1.5x upper limit of normal range at the investigator site
   * Aspartate aminotransferase (AST) and / or alanine aminotransferase (ALT) less than or equal to 1.5x upper limit of normal range at the investigator site (It is the same if patients have liver metastases)
   * PaO2 or SpO2 more than 60torr or 92%
7. Written informed consent that is consistent with ICH-GCP guidelines.

Exclusion criteria:

1. Patients who have received chemotherapy (including other investigational drug), hormonal therapy and immune therapy =<4 weeks prior to registration or who have not recovered from side effects of such therapy.
2. Patients who have received radiotherapy =<4 weeks (limited field (e.g brain or bone metastasis) radiation =<2 weeks) prior to registration.
3. Patients who have active brain metastases. (Patients who have no symptoms and is not needed to receive therapy in the registration may participate in this trial)
4. Patients with active double cancer. (Patients who have skin cancer that is not malignant melanoma and carcinoma in situ of uterine cervix may participate in this trial)
5. Patients with distinct / suspected pulmonary fibrosis or interstitial lung disease by the chest radiographic findings, or patients with a previous history of.
6. History of clinically significant haemoptysis within the past 3 months (more than one tea spoon of fresh blood per day)
7. Therapeutic anticoagulation (except low dose heparin and/or heparin flush as needed for maintenance of an indwelling intravenous device) or antiplatelet therapy (except for chronic low-dose therapy with acetylsalicylic acid =<325 mg per day)
8. History of major thrombotic or clinically relevant major bleeding event in the past 6 months prior to registration.
9. Known inherited predisposition to bleeding or thrombosis.
10. Significant cardiovascular diseases. (i.e. hypertension not controlled by medical therapy, unstable angina, history of myocardial infarction within the past 6 months, congestive heart failure > NYHA II, serious cardiac arrhythmia, pericardial effusion)
11. Significant weight loss (> 10 %) within the past 6 weeks prior to registration in the this trial
12. Current peripheral neuropathy >= CTCAE grade 2 except due to trauma.
13. Accumulation of coelomic fluid (e.g. pleural effusion, ascites fluid, cardiac effusion) requiring treatment
14. Major injuries and/or surgery within the past 10 days prior to registration with incomplete wound healing.
15. Serious infections requiring systemic antibiotic (e.g antiviral, antimicrobial, antifungal) therapy.
16. Decompensated diabetes mellitus or other contraindication to high dose corticosteroid therapy.
17. Gastrointestinal disorders or abnormalities (e.g Crohn's disease, Colitis ulcerosa and extensive gastrectomy) that would interfere with absorption of the study drug.
18. Patients with difficulty in swallowing study medication
19. Patients with positive HBs antigen, HCV antibody, or HIV antibody test
20. Serious illness or concomitant non-oncological disease such as neurologic-, psychiatric-, infectious disease or active ulcers (gastro-intestinal tract, skin) or laboratory abnormality that may increase the risk associated with trial participation or investigational drug administration and in the judgment of the investigator would make the patient inappropriate for entry into the trial.
21. Patients who are sexually active and unwilling to use a medically acceptable method of contraception (e.g. such as implants, injectables, combined oral contraceptives, some intrauterine devices or vasectomized partner for participating females, condoms for participating males) during the trial and for at least 12 months after end of active therapy
22. Female patients who are pregnant, breast feeding and may become pregnant.
23. Patients who have or is suspected of having active alcohol or drug abuse.
24. Patient with clinically meaningful drug hypersensitivities.
25. Patients with auto immune disease.
26. Patients unable to comply with the protocol.
27. Other patients judged ineligible for enrolment in the study by the investigator.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-03; Primary Completion 2012-09 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (2):
- Japan (2):
  - 1199.29.002 Boehringer Ingelheim Investigational Site, Fukuoka, Fukuoka
  - 1199.29.001 Boehringer Ingelheim Investigational Site, Osaka-Sayamashi, Osaka

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 43 patients entered.1 patient was replaced because he did not take any nintedanib(Nin) due to new brain metastasis after completion of first administration of docetaxel. Accordingly,42 patients treated with at least 1 dose of Nin in combination with docetaxel.Patients started mono therapy phase after discontinued from combination therapy phase .
Pre-assignment Details: In case a patient had to discontinue docetaxel for reasons other than progression disease, the patient could continue therapy with nintedanib if the patient had been treated with combination therapy with docetaxel during at least 4 treatment courses.
Groups:
- Nintedanib 100 mg + Docetaxel 60 mg/m2: Patients administered a soft gelatin capsule of nintedanib 100 mg, orally, twice daily (b.i.d.) from day 2 in combination with docetaxel 60 mg/m2 injection once every three weeks administered via intravenous infusion over one hour. Nintedanib was not taken when docetaxel was administered.
- Nintedanib 150 mg + Docetaxel 60 mg/m2 (BSA <1.5 m^2): Patients with body surface area (BSA) <1.5 m^2 administered a soft gelatin capsule of nintedanib 150 mg, orally, b.i.d. from day 2 in combination with docetaxel 60 mg/m2, injection once every three weeks administered via intravenous infusion over one hour. Nintedanib was not taken when docetaxel was administered.
- Nintedanib 150 mg + Docetaxel 60 mg/m2 (BSA >=1.5 m^2): Patients with body surface area ≥1.5 m^2 administered a soft gelatin capsule of nintedanib 150 mg, orally, b.i.d. from day 2 in combination with docetaxel 60 mg/m2, injection once every three weeks administered via intravenous infusion over one hour. Nintedanib was not taken when docetaxel was administered.
- Nintedanib 150 mg + Docetaxel 75 mg/m2 (BSA <1.5 m^2): Patients with body surface area <1.5 m^2 administered a soft gelatin capsule of nintedanib 150 mg, orally, b.i.d. from day 2 in combination with docetaxel 75 mg/m2 injection once every three weeks administered via intravenous infusion over one hour. Nintedanib was not taken when docetaxel was administered.
- Nintedanib 150 mg + Docetaxel 75 mg/m2 (BSA >=1.5 m^2): Patients with body surface area ≥1.5 m^2 administered a soft gelatin capsule of nintedanib 150 mg, orally, b.i.d. from day 2 in combination with docetaxel 75 mg/m2 injection once every three weeks administered via intravenous infusion over one hour. Nintedanib was not taken when docetaxel was administered.
- Nintedanib 200 mg + Docetaxel 60 mg/m2 (BSA <1.5 m^2): Patients with body surface area <1.5 m^2 administered a soft gelatin capsule of nintedanib 200 mg, orally, b.i.d. from day 2 in combination with docetaxel 60 mg/m2 injection once every three weeks administered via intravenous infusion over one hour. Nintedanib was not taken when docetaxel was administered.
- Nintedanib 200 mg + Docetaxel 60 mg/m2 (BSA >=1.5 m^2): Patients with body surface area ≥1.5 m^2 administered a soft gelatin capsule of nintedanib 200 mg, orally, b.i.d. from day 2 in combination with docetaxel 60 mg/m2 injection once every three weeks administered via intravenous infusion over one hour. Nintedanib was not taken when docetaxel was administered.
- Nintedanib 200 mg + Docetaxel 75 mg/m2 (BSA >=1.5 m^2): Patients with body surface area ≥1.5 m^2 administered a soft gelatin capsule of nintedanib 200 mg, orally, b.i.d. from day 2 in combination with docetaxel 75 mg/m2 injection once every three weeks administered via intravenous infusion over one hour. Nintedanib was not taken when docetaxel was administered.
Period: Combination Therapy Phase
Arm/Group | Nintedanib 100 mg + Docetaxel 60 mg/m2 | Nintedanib 150 mg + Docetaxel 60 mg/m2 (BSA <1.5 m^2) | Nintedanib 150 mg + Docetaxel 60 mg/m2 (BSA >=1.5 m^2) | Nintedanib 150 mg + Docetaxel 75 mg/m2 (BSA <1.5 m^2) | Nintedanib 150 mg + Docetaxel 75 mg/m2 (BSA >=1.5 m^2) | Nintedanib 200 mg + Docetaxel 60 mg/m2 (BSA <1.5 m^2) | Nintedanib 200 mg + Docetaxel 60 mg/m2 (BSA >=1.5 m^2) | Nintedanib 200 mg + Docetaxel 75 mg/m2 (BSA >=1.5 m^2)
Started | 3 | 7 | 3 | 6 | 7 | 3 | 8 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 7 | 3 | 6 | 7 | 3 | 8 | 6
Not completed — Progressive disease | 2 | 3 | 3 | 3 | 3 | 1 | 1 | 1
Not completed — Dose limiting toxicity | 0 | 1 | 0 | 1 | 1 | 2 | 2 | 1
Not completed — Adverse Event | 0 | 2 | 0 | 2 | 2 | 0 | 3 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other reason not defined above | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Not treated | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Mono Therapy Phase
Arm/Group | Nintedanib 100 mg + Docetaxel 60 mg/m2 | Nintedanib 150 mg + Docetaxel 60 mg/m2 (BSA <1.5 m^2) | Nintedanib 150 mg + Docetaxel 60 mg/m2 (BSA >=1.5 m^2) | Nintedanib 150 mg + Docetaxel 75 mg/m2 (BSA <1.5 m^2) | Nintedanib 150 mg + Docetaxel 75 mg/m2 (BSA >=1.5 m^2) | Nintedanib 200 mg + Docetaxel 60 mg/m2 (BSA <1.5 m^2) | Nintedanib 200 mg + Docetaxel 60 mg/m2 (BSA >=1.5 m^2) | Nintedanib 200 mg + Docetaxel 75 mg/m2 (BSA >=1.5 m^2)
Started | 0 | 1 (One patient started mono therapy phase after discontinued from combination therapy phase.) | 0 | 1 (One patient started mono therapy phase after discontinued from combination therapy phase.) | 2 (Two patients started mono therapy phase after discontinued from combination therapy phase.) | 0 | 1 (One patient started mono therapy phase after discontinued from combination therapy phase.) | 3 (Three patients started mono therapy phase after discontinued from combination therapy phase.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 3
Not completed — Progressive disease | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set: all patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Nintedanib 100 mg + Docetaxel 60 mg/m2 | Nintedanib 150 mg + Docetaxel 60 mg/m2 (BSA <1.5 m^2) | Nintedanib 150 mg + Docetaxel 60 mg/m2 (BSA >=1.5 m^2) | Nintedanib 150 mg + Docetaxel 75 mg/m2 (BSA <1.5 m^2) | Nintedanib 150 mg + Docetaxel 75 mg/m2 (BSA >=1.5 m^2) | Nintedanib 200 mg + Docetaxel 60 mg/m2 (BSA <1.5 m^2) | Nintedanib 200 mg + Docetaxel 60 mg/m2 (BSA >=1.5 m^2) | Nintedanib 200 mg + Docetaxel 75 mg/m2 (BSA >=1.5 m^2) | Total
Number analyzed (Participants) | 3 | 7 | 3 | 6 | 7 | 3 | 7 | 6 | 42
Age, Continuous [Median (Full Range); unit: years] | 58.0 [49 to 58] | 68.0 [59 to 71] | 64.0 [60 to 69] | 65.0 [45 to 70] | 63.0 [60 to 73] | 62.0 [58 to 72] | 64.0 [47 to 72] | 61.5 [51 to 72] | 63.5 [45 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 0 | 4 | 1 | 3 | 1 | 0 | 13
  Male | 2 | 4 | 3 | 2 | 6 | 0 | 6 | 6 | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Dose Limited Toxicity in Combination Therapy of Nintedanib and Docetaxel
Description: Number of participants experienced Dose Limited Toxicity (DLT) in combination therapy of nintedanib and docetaxel.
  Maximum tolerated dose (MTD) of nintedanib combination with docetaxel were to be determined separately in the patient groups of body surface area (BSA) <1.5 m2 and BSA ≥1.5 m2. The MTD were to be determined as a combination of a dose equal to or less than 200 mg b.i.d. of nintedanib and 60 mg/m2 and 75 mg/m2 every 3 weeks of docetaxel at which either 0 out of 3, 1 out of 6, or 2 out of 6 patients experienced DLT.
Time Frame: During the first treatment course, up to 3 weeks
Population: Treated set (Patients eligible for DLT confirmation)
Measure: Number; unit: Participants
Arm/Group | Nintedanib 100 mg + Docetaxel 60 mg/m2 | Nintedanib 150 mg + Docetaxel 60 mg/m2 (BSA <1.5 m^2) | Nintedanib 150 mg + Docetaxel 60 mg/m2 (BSA >=1.5 m^2) | Nintedanib 150 mg + Docetaxel 75 mg/m2 (BSA <1.5 m^2) | Nintedanib 150 mg + Docetaxel 75 mg/m2 (BSA >=1.5 m^2) | Nintedanib 200 mg + Docetaxel 60 mg/m2 (BSA <1.5 m^2) | Nintedanib 200 mg + Docetaxel 60 mg/m2 (BSA >=1.5 m^2) | Nintedanib 200 mg + Docetaxel 75 mg/m2 (BSA >=1.5 m^2)
Number analyzed (Participants) | 3 | 6 | 3 | 6 | 6 | 3 | 6 | 6
Participants | 0 | 2 | 0 | 1 | 2 | 3 | 2 | 2

2. Primary Outcome: Adverse Events According to Common Terminology Criteria for Adverse Events (CTCAE), Version 3.0 for All Courses
Description: Number of participants with adverse events according to Common Terminology Criteria for Adverse Events (CTCAE), version 3.0 for all courses.
  The CTCAE grades are: 1 (mild AE), 2 (moderate AE), 3 (severe AE), 4 (life-threatening or disabling AE), 5 (death related to AE).
Time Frame: Between the first administration of docetaxel and 28 days after last administration of docetaxel and/or nintedanib, up to 1367 days
Population: Treated set
Measure: Number; unit: Participants
Arm/Group | Nintedanib 100 mg + Docetaxel 60 mg/m2 | Nintedanib 150 mg + Docetaxel 60 mg/m2 (BSA <1.5 m^2) | Nintedanib 150 mg + Docetaxel 60 mg/m2 (BSA >=1.5 m^2) | Nintedanib 150 mg + Docetaxel 75 mg/m2 (BSA <1.5 m^2) | Nintedanib 150 mg + Docetaxel 75 mg/m2 (BSA >=1.5 m^2) | Nintedanib 200 mg + Docetaxel 60 mg/m2 (BSA <1.5 m^2) | Nintedanib 200 mg + Docetaxel 60 mg/m2 (BSA >=1.5 m^2) | Nintedanib 200 mg + Docetaxel 75 mg/m2 (BSA >=1.5 m^2)
Number analyzed (Participants) | 3 | 7 | 3 | 6 | 7 | 3 | 7 | 6
Participants
  Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0
  Grade 4 | 3 | 6 | 1 | 5 | 7 | 3 | 5 | 6
  Grade 5 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0

3. Secondary Outcome: Objective Tumor Response
Description: Number of participants with objective response defined as complete response (CR) or partial response (PR) according to the Response Evaluation Criteria In Solid Tumors (RECIST) version 1.0
Time Frame: Pre-treatment, every 6 weeks from treatment course 3, end of treatment (up to 1367 days)
Population: Patients who were treated with nintedanib and had both baseline and at least one post-treatment tumour measurement by computed tomography (CT) image
Measure: Number; unit: Participants
Groups:
- Nintedanib 150 mg + Docetaxel 60 mg/m2: Patients administered a soft gelatin capsule of nintedanib 150 mg, orally, twice daily (b.i.d.) from day 2 in combination with docetaxel 60 mg/m2 injection once every three weeks administered via intravenous infusion over one hour. Nintedanib was not taken when docetaxel was administered.
- Nintedanib 150 mg + Docetaxel 75 mg/m2: Patients administered a soft gelatin capsule of nintedanib 150 mg, orally, twice daily (b.i.d.) from day 2 in combination with docetaxel 75 mg/m2 injection once every three weeks administered via intravenous infusion over one hour. Nintedanib was not taken when docetaxel was administered.
- Nintedanib 200 mg + Docetaxel 60 mg/m2: Patients administered a soft gelatin capsule of nintedanib 200 mg, orally, twice daily (b.i.d.) from day 2 in combination with docetaxel 60 mg/m2 injection once every three weeks administered via intravenous infusion over one hour. Nintedanib was not taken when docetaxel was administered.
- Nintedanib 200 mg + Docetaxel 75 mg/m2: Patients administered a soft gelatin capsule of nintedanib 200 mg, orally, twice daily (b.i.d.) from day 2 in combination with docetaxel 75 mg/m2 injection once every three weeks administered via intravenous infusion over one hour. Nintedanib was not taken when docetaxel was administered.
Arm/Group | Nintedanib 100 mg + Docetaxel 60 mg/m2 | Nintedanib 150 mg + Docetaxel 60 mg/m2 | Nintedanib 150 mg + Docetaxel 75 mg/m2 | Nintedanib 200 mg + Docetaxel 60 mg/m2 | Nintedanib 200 mg + Docetaxel 75 mg/m2
Number analyzed (Participants) | 3 | 9 | 12 | 8 | 6
Participants
  Yes | 0 | 2 | 5 | 2 | 1
  No | 3 | 7 | 7 | 6 | 5

4. Secondary Outcome: Disease Control
Description: Number of participants with disease control, defined as complete response (CR) or partial response (PR) or stable disease (SD) according to the Response Evaluation Criteria In Solid Tumors (RECIST) 1.0
Time Frame: Pre-treatment, every 6 weeks from treatment course 3, end of treatment (up to 1367 days)
Population: Patients who treated with nintedanib and had both baseline and at least one post-treated tumour measurement by computed tomography (CT) image
Measure: Number; unit: Participants
Arm/Group | Nintedanib 100 mg + Docetaxel 60 mg/m2 | Nintedanib 150 mg + Docetaxel 60 mg/m2 | Nintedanib 150 mg + Docetaxel 75 mg/m2 | Nintedanib 200 mg + Docetaxel 60 mg/m2 | Nintedanib 200 mg + Docetaxel 75 mg/m2
Number analyzed (Participants) | 3 | 9 | 12 | 8 | 6
Participants
  Yes | 2 | 5 | 12 | 5 | 4
  No | 1 | 4 | 0 | 3 | 2

5. Secondary Outcome: Progression-Free Survival (PFS)
Description: For participants with known date of progression or death (of any cause): PFS [days] = earlier of date of progression or death - date the study treatment started + 1.
  For participants known to be alive without progression by the end of trial or follow-up visit: PFS (censored) [days] = date of last imaging when the participant is known to be progression-free and alive - date the study treatment started + 1.
  Progression is assessed according to RECIST version 1.0.
Time Frame: Pre-treatment, every 6 weeks from treatment course 3, end of treatment (up to 1367 days)
Population: Treated set
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Nintedanib 100 mg + Docetaxel 60 mg/m2 | Nintedanib 150 mg + Docetaxel 60 mg/m2 | Nintedanib 150 mg + Docetaxel 75 mg/m2 | Nintedanib 200 mg + Docetaxel 60 mg/m2 | Nintedanib 200 mg + Docetaxel 75 mg/m2
Number analyzed (Participants) | 3 | 10 | 13 | 10 | 6
Days | 229.5 [200.0 to 259.0] | 117.0 [36.0 to 267.0] | 139.0 [87.0 to 262.0] | 351.0 [131.0 to 614.0] | 184.0 [68.0 to 884.0]

6. Secondary Outcome: Time to Treatment Failure (TTF)
Description: For participants with known date of discontinuation of the study treatment (or progression [not necessarily confirmed by tumour imaging; can also be based on any clinical sign of tumour progression] or death): TTF [days] = earlier of date of discontinuation of the study treatment, progression, or death - date the study treatment started + 1.
  For participants known to be alive without progression by the end of trial or follow-up visit: TTF (censored) [days] = date when the patient is known to be progression-free and alive - date the study treatment started + 1.
  Progression is assessed according to RECIST version 1.0.
Time Frame: Pre-treatment, every 6 weeks from treatment course 3, end of treatment (up to 1367 days)
Population: Treated set
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Nintedanib 100 mg + Docetaxel 60 mg/m2 | Nintedanib 150 mg + Docetaxel 60 mg/m2 | Nintedanib 150 mg + Docetaxel 75 mg/m2 | Nintedanib 200 mg + Docetaxel 60 mg/m2 | Nintedanib 200 mg + Docetaxel 75 mg/m2
Number analyzed (Participants) | 3 | 10 | 13 | 10 | 6
Days | 200.0 [54.0 to 259.0] | 83.5 [10.0 to 187.0] | 134.0 [75.0 to 178.0] | 87.0 [8.0 to 212.0] | 176.0 [52.0 to 884.0]

7. Secondary Outcome: Clinical Relevant Abnormalities in Laboratory Parameters
Description: Number of participants with clinically relevant abnormalities in laboratory parameters reported as adverse events
Time Frame: as for outcome 2
Population: Treated set
Measure: Number; unit: Participants
Arm/Group | Nintedanib 100 mg + Docetaxel 60 mg/m2 | Nintedanib 150 mg + Docetaxel 60 mg/m2 (BSA <1.5 m^2) | Nintedanib 150 mg + Docetaxel 60 mg/m2 (BSA >=1.5 m^2) | Nintedanib 150 mg + Docetaxel 75 mg/m2 (BSA <1.5 m^2) | Nintedanib 150 mg + Docetaxel 75 mg/m2 (BSA >=1.5 m^2) | Nintedanib 200 mg + Docetaxel 60 mg/m2 (BSA <1.5 m^2) | Nintedanib 200 mg + Docetaxel 60 mg/m2 (BSA >=1.5 m^2) | Nintedanib 200 mg + Docetaxel 75 mg/m2 (BSA >=1.5 m^2)
Number analyzed (Participants) | 3 | 7 | 3 | 6 | 7 | 3 | 7 | 6
Participants
  Alanine aminotransferase increased | 2 | 4 | 0 | 5 | 4 | 3 | 4 | 5
  Aspartate aminotransferase increased | 2 | 4 | 0 | 5 | 4 | 3 | 4 | 5
  Blood alkaline phosphatase increased | 0 | 3 | 0 | 4 | 4 | 3 | 2 | 3
  Gamma-glutamyltransferase increased | 1 | 4 | 0 | 4 | 4 | 3 | 4 | 4
  Blood bilirubin increased | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0
  Platelet count decreased | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
  White blood cell count decreased | 0 | 1 | 0 | 3 | 2 | 0 | 0 | 2
  Blood calcium decreased | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
  Gamma-glutamyltransferase | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
  Blood chloride decreased | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Blood thyroid stimulating hormone increased | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
  Blood urea increased | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  C-reactive protein increased | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1
  Haemoglobin decreased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Lymphocyte count decreased | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Neutrophil count decreased | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
  Prothrombin level decreased | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Tri-iodothyronine free decreased | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Blood albumin decreased | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Blood potassium decreased | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Blood uric acid increased | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Blood urine | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Blood urine present | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Electrocardiogram QT prolonged | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: AUC0-inf of Nintedanib in Course 1
Description: AUC0-inf (area under the plasma concentration-time curve over the time interval from 0 extrapolated to infinity) after the first administration of nintedanib in course 1
Time Frame: -0:05 hours (h) before drug administration and 1h, 2h, 3h, 4h, 6h, 7h, 10h and 23:55h after drug administration in course 1
Population: Treated set (AUC0-inf could not be calculated in 5 patients because the elimination phase was not observed in plasma concentration-time profiles in these patients.)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Nintedanib 100 mg: Patients with Nintedanib 100 mg b.i.d.
- Nintedanib 150 mg: Patients with Nintedanib 150 mg b.i.d.
- Nintedanib 200 mg: Patients with Nintedanib 200 mg b.i.d.
Arm/Group | Nintedanib 100 mg | Nintedanib 150 mg | Nintedanib 200 mg
Number analyzed (Participants) | 3 | 18 | 16
ng*h/mL | 169 (56.1) | 260 (50.1) | 349 (25.6)

9. Secondary Outcome: Cmax of Nintedanib in Course 1
Description: Cmax (maximum measured plasma concentration) after the first administration of nintedanib in course 1
Time Frame: -0:05h before drug administration and 1h, 2h, 3h, 4h, 6h, 7h, 10h and 23:55h after drug administration in course 1
Population: Treated set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Nintedanib 100 mg | Nintedanib 150 mg | Nintedanib 200 mg
Number analyzed (Participants) | 3 | 23 | 16
ng/mL | 29.3 (60.0) | 33.4 (91.1) | 59.9 (43.9)

10. Secondary Outcome: AUC0-inf of Docetaxel in Course 1
Description: AUC0-inf (area under the plasma concentration-time curve over the time interval from 0 extrapolated to infinity) after the first administration of docetaxel in course 1
Time Frame: -0:05h before drug administration and 1h, 1.5h, 2h, 3h, 4h, 7h, 23:55h and 47:55h after drug administration
Population: Treated set (1 patient was replaced after completion of first administration of docetaxel and before any nintedanib intake. Pharmacokinetic (PK) sampling of docetaxel for this patient was done and included in PK analysis.)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Docetaxel 60 mg/m2: Patients with Docetaxel 60 mg/m2
- Docetaxel 75 mg/m2: Patients with Docetaxel 75 mg/m2
Arm/Group | Docetaxel 60 mg/m2 | Docetaxel 75 mg/m2
Number analyzed (Participants) | 24 | 19
ng*h/mL | 3270 (35.6) | 3810 (22.7)

11. Secondary Outcome: Cmax of Docetaxel in Course 1
Description: Cmax (maximum measured plasma concentration) after the first administration of docetaxel in course 1
Time Frame: -0:05h before drug administration and 1h, 1.5h, 2h, 3h, 4h, 7h, 23:55h and 47:55h after drug administration
Population: Treated set (1 patient was replaced after completion of first administration of docetaxel and before any nintedanib intake. PK sampling of docetaxel for this patient was done and included in PK analysis.)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Docetaxel 60 mg/m2 | Docetaxel 75 mg/m2
Number analyzed (Participants) | 24 | 19
ng/mL | 3150 (42.8) | 3550 (32.2)

12. Secondary Outcome: AUC0-inf of Docetaxel in Course 2
Description: AUC0-inf (area under the plasma concentration-time curve over the time interval from 0 extrapolated to infinity) after the first administration of docetaxel in course 2.
  Docetaxel 50 mg/m2 patients were assigned to Docetaxel 60 mg/m2 in Cycle 1, but the dose was reduced to 50 mg/m2 in Cycle 2 as defined in the Clinical Trial Protocol.
Time Frame: -0:05h before drug administration and 1h, 1.5h, 2h, 3h, 4h, 7h, 23:55h and 47:55h after drug administration
Population: Treated set (AUC0-inf could not be calculated in 1 patient because the elimination phase was not observed in plasma concentration-time profile in this patient.)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Docetaxel 50 mg/m2: Patients with Docetaxel 50 mg/m2
Arm/Group | Docetaxel 50 mg/m2 | Docetaxel 60 mg/m2 | Docetaxel 75 mg/m2
Number analyzed (Participants) | 2 | 16 | 8
ng*h/mL | 2320 (14.9) | 3750 (31.1) | 4270 (34.2)

13. Secondary Outcome: Cmax of Docetaxel in Course 2
Description: Cmax (maximum measured plasma concentration) after the first administration of docetaxel in course 2.
  Docetaxel 50 mg/m2 patients were assigned to Docetaxel 60 mg/m2 in Cycle 1, but the dose was reduced to 50 mg/m2 in Cycle 2 as defined in the Clinical Trial Protocol.
Time Frame: -0:05h before drug administration and 1h, 1.5h, 2h, 3h, 4h, 7h, 23:55h and 47:55h after drug administration
Population: Treated set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Docetaxel 50 mg/m2 | Docetaxel 60 mg/m2 | Docetaxel 75 mg/m2
Number analyzed (Participants) | 2 | 16 | 9
ng/mL | 1870 (33.9) | 3740 (33.7) | 4070 (56.7)

ADVERSE EVENTS:
Time Frame: between the first administration of docetaxel and 28 days after last administration of docetaxel and/or nintedanib, up to 1367 days
Arm/Group | Nintedanib 100 mg + Docetaxel 60 mg/m2 | Nintedanib 150 mg + Docetaxel 60 mg/m2 (BSA <1.5 m^2) | Nintedanib 150 mg + Docetaxel 60 mg/m2 (BSA >=1.5 m^2) | Nintedanib 150 mg + Docetaxel 75 mg/m2 (BSA <1.5 m^2) | Nintedanib 150 mg + Docetaxel 75 mg/m2 (BSA >=1.5 m^2) | Nintedanib 200 mg + Docetaxel 60 mg/m2 (BSA <1.5 m^2) | Nintedanib 200 mg + Docetaxel 60 mg/m2 (BSA >=1.5 m^2) | Nintedanib 200 mg + Docetaxel 75 mg/m2 (BSA >=1.5 m^2)
Serious Adverse Events (participants affected / at risk) | 1/3 | 4/7 | 0/3 | 2/6 | 4/7 | 0/3 | 3/7 | 1/6
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 3/3 | 6/6 | 7/7 | 3/3 | 7/7 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib 100 mg + Docetaxel 60 mg/m2 (N=3) | Nintedanib 150 mg + Docetaxel 60 mg/m2 (BSA <1.5 m^2) (N=7) | Nintedanib 150 mg + Docetaxel 60 mg/m2 (BSA >=1.5 m^2) (N=3) | Nintedanib 150 mg + Docetaxel 75 mg/m2 (BSA <1.5 m^2) (N=6) | Nintedanib 150 mg + Docetaxel 75 mg/m2 (BSA >=1.5 m^2) (N=7) | Nintedanib 200 mg + Docetaxel 60 mg/m2 (BSA <1.5 m^2) (N=3) | Nintedanib 200 mg + Docetaxel 60 mg/m2 (BSA >=1.5 m^2) (N=7) | Nintedanib 200 mg + Docetaxel 75 mg/m2 (BSA >=1.5 m^2) (N=6)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peritumoural oedema (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib 100 mg + Docetaxel 60 mg/m2 (N=3) | Nintedanib 150 mg + Docetaxel 60 mg/m2 (BSA <1.5 m^2) (N=7) | Nintedanib 150 mg + Docetaxel 60 mg/m2 (BSA >=1.5 m^2) (N=3) | Nintedanib 150 mg + Docetaxel 75 mg/m2 (BSA <1.5 m^2) (N=6) | Nintedanib 150 mg + Docetaxel 75 mg/m2 (BSA >=1.5 m^2) (N=7) | Nintedanib 200 mg + Docetaxel 60 mg/m2 (BSA <1.5 m^2) (N=3) | Nintedanib 200 mg + Docetaxel 60 mg/m2 (BSA >=1.5 m^2) (N=7) | Nintedanib 200 mg + Docetaxel 75 mg/m2 (BSA >=1.5 m^2) (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 4 | 2 | 0 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 3 | 7 | 1 | 3 | 6 | 3 | 7 | 5
Lymphopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 3 | 1 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 7 | 2 | 6 | 7 | 3 | 7 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 1 | 1 | 3 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye discharge (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1 | 1 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 3
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 1 | 2 | 0 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 4 | 1 | 2 | 6 | 2 | 4 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 5 | 0 | 2 | 1 | 1 | 2 | 3
Periodontal disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 3 | 1 | 1 | 1 | 0 | 3 | 3
Tongue discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 5 | 0 | 3 | 3 | 1 | 1 | 1
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 7 | 1 | 6 | 5 | 2 | 4 | 6
Influenza like illness (General disorders) | 1 | 0 | 0 | 1 | 3 | 0 | 1 | 1
Injection site reaction (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Oedema (General disorders) | 2 | 2 | 0 | 2 | 1 | 0 | 0 | 2
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 4 | 2 | 1 | 1 | 4
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Eyelid infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1
Infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Nail infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 2
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Oral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulpitis dental (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 4 | 0 | 5 | 4 | 3 | 4 | 5
Aspartate aminotransferase increased (Investigations) | 2 | 4 | 0 | 5 | 4 | 3 | 4 | 5
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 3 | 0 | 4 | 4 | 3 | 2 | 3
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0
Blood calcium decreased (Investigations) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Blood chloride decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Blood urea increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood urine (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood urine present (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 1 | 4 | 0 | 4 | 4 | 3 | 4 | 4
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Prothrombin level decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tri-iodothyronine free decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 2
Weight increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 3 | 2 | 0 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 2 | 5 | 2 | 6 | 3 | 3 | 6 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hypovitaminosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 2 | 0 | 1 | 3 | 3 | 3 | 4
Headache (Nervous system disorders) | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 0 | 0 | 2 | 3 | 0 | 1 | 2
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Visual field defect (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 2
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 4 | 0 | 6 | 6 | 1 | 4 | 6
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nail bed bleeding (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 1 | 2 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 2 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 4 | 3 | 1 | 3 | 3
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin swelling (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vasculitis (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.